CLINICAL TRIAL: NCT04274504
Title: Osteopontin Level and Promoter Polymorphism in Egyptian Metastatic Breast Cancer Patients
Brief Title: Osteopontin in Metastatic Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 2019035
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Survival, Prosthesis
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — The PCR amplification of the promoter regulatory region from the extracted DNA by using the following primers -3 (forward primer 5" -CAA GCT ACT GCA TAC TCG AAA TCA CA-3" ; reverse primer 5" - ACA ACC AAG CCC TCC CAG AAT TTA-3" ). PCR was performed using 50 ng DNA as a template under the following conditions: 95°C for 10 min, then 36 cycles of 94°C for 30 s, an annealing temperature for 60 s, and 72°C for 60 s, with a final extension at 72°C for 15 min. After affinity membrane purification using the QIAquick Gel Extraction kit (Qiagen, Carlsbad, CA, USA), the PCR products were subjected to cycle sequencing with the respective forward and reverse primer using an automated ABI 310 DNA sequencer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: metatstatic breast
  Interventions: Diagnostic Test: Osteopontin

INTERVENTIONS:
Diagnostic Test: Osteopontin — Serum osteopontin (OPN) was measured by ELIZA and osteopontin gene mutation was analyzed by sequencing and correlated with clinicopathological criteria, response, PFS and OS.

SUMMARY:
OPN plays an important role in various aspects of malignancy, particularly those involved in tissue invasion and metastasis, and OPN levels have been associated with aggressive¬ness in several cancer types, including breast cancer. Tumor response to treatment is a predictor of prognosis and overall survival for cancer patient population the investigators assigned osteopontin as potential contributors in breast cancer.

DETAILED DESCRIPTION:
Analysis of polymorphisms in the OPN regulatory region:

The PCR amplification of the promoter regulatory region from the extracted DNA by using the following primers -3 (forward primer 5" -CAA GCT ACT GCA TAC TCG AAA TCA CA-3" ; reverse primer 5" - ACA ACC AAG CCC TCC CAG AAT TTA-3" ). PCR was performed using 50 ng DNA as a template under the following conditions: 95°C for 10 min, then 36 cycles of 94°C for 30 s, an annealing temperature for 60 s, and 72°C for 60 s, with a final extension at 72°C for 15 min. After affinity membrane purification using the QIAquick Gel Extraction kit (Qiagen, Carlsbad, CA, USA), the PCR products were subjected to cycle sequencing with the respective forward and reverse primer using an automated ABI 310 DNA sequencer.

Measurement of serum level of osteopontin:

OPN level were measured using Enzyme linked immnosorbent (ELISA) Kit supplied by IBL (Immuno-Biological laboratories Co. Ltd., Japan). 30 normal females were conducted with matched age with a median osteopontine serum level of 15 so, this level was assigned as a cut off value.

Pretreatment serum level and polymorphism of oteopontine was correlated with different clinicopathological criteria of the patients, response to the treatment, PFS and OS.

ELIGIBILITY:
Inclusion Criteria:

* de novo metastatic breast cancer patients recruited from Oncology center Mansoura University and clinical oncology department, Mansoura University Hospital All included patients were presented with disseminated visceral +/- bone metastasis (visceral crisis)

Exclusion Criteria:

* brain metastasis was excluded

Ages: 31 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Denovo Metastatic breast
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Both pretreatment serum level of oteopontin and gene mutation were correlated with different clinicopathological criteria of the patients, response to the treatment, PFS and OS. | 2 years
  Serum osteopontin (OPN) was measured by ELIZA and osteopontin gene mutation was analyzed by sequencing and correlated with clinicopathological criteria, response, PFS and OS.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Elbaiomy, Principal Investigator — Mansoura university Oncology Center
Locations (1):
- Mansoura University Oncology Center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No